CLINICAL TRIAL: NCT02585752
Title: A Study of Expiratory Pressure Modulation in Moderate to Severe COPD Patients - Phase 1b
Acronym: ComfortCOPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-177 / AA-CmfCOPD-02
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Single centre, single arm (Experimental): Noninvasive ventilation with expiratory modulation. Assessment of comfort and blood gases.
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: Noninvasive ventilation — Expiratory pressure modulation

SUMMARY:
Dynamic pulmonary hyperinflation (DH) and intrinsic positive end-expiratory pressure (PEEP) are well known problems in COPD patients with acute and chronic respiratory failure. Measurement of intrinsic PEEP level during both, invasive and non-invasive ventilation is of major importance since in some circumstances (e.g. during exercise or during exacerbations) it can significantly increase respiratory workload of COPD patients. Extrinsic PEEP applied during both, invasive and noninvasive ventilation is used to overcome intrinsic PEEP and therefore to avoid or reduce dynamic hyperinflation.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years who are contractually capable and mentally able to understand and follow the instructions of the study personnel
2. Signed informed consent
3. Moderate to severe COPD patients (FEV1/FVC ratio <70% and FEV1 < 50% pred) with chronic hypercapnic respiratory failure (PaCO2 >45 mmHg)
4. Currently using NIV

Exclusion Criteria:

1. Acute exacerbation of COPD, acute respiratory failure (ph < 7,35 and/or respiratory rate >30/min)
2. Unstable heart failure
3. Cardiac failure with dehydration
4. Pregnancy/breastfeeding women
5. Pneumothorax/-mediastinum
6. Increased risk of pneumothorax, pneumomediastinum or venous air embolism
7. In the opinion of the investigator, the patient is unsuitable for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 day
  Subjective rating of comfort during expiration

SECONDARY OUTCOMES:
Minute ventilation | 1 day
  Volume of inhaled air in one minute (L/min)
Respiratory rate | 1 day
  Number of breaths per minute (breaths/min)
Tidal volume | 1 day
  Volume of air that is inhaled or exhaled during normal breathing (mL)
CO2 transcutaneous (tcCO2) | 1 day
  Arterial carbon dioxide partial pressure (mm Hg)
pO2 arterial (paO2) | 1 day
  Arterial oxygen partial pressure (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, MD, Principal Investigator — Universitätsklinikum Aachen
Locations (1):
- Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Cornelissen CG, Müller T, Schmitz S, Dreher M. Nichtinvasive Beatmung: Patientenkomfort und Sicherheit einer Modulation des expiratorischen Flusses. Pneumologie 2018; 72(S01), S11